CLINICAL TRIAL: NCT01387555
Title: A Phase 2b Randomized Trial of JX-594 (Vaccinia GM-CSF / TK-deactivated Virus) Plus Best Supportive Care Versus Best Supportive Care in Patients With Advanced Hepatocellular Carcinoma Who Have Failed Sorafenib Treatment
Brief Title: A Phase 2b Study of Modified Vaccinia Virus to Treat Patients Advanced Liver Cancer Who Failed Sorafenib
Acronym: TRAVERSE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jennerex Biotherapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JX594-HEP018
Record Dates: First submitted 2011-06-27; First posted 2011-07-04 (Estimated); Last update posted 2015-03-11 (Estimated); Status verified 2015-03

CONDITIONS: Hepatocellular Carcinoma; Liver Cancer; HCC
Keywords: liver cancer; liver tumor; advanced hcc; hepatocellular cancer; Jennerex; HCC; sorafenib; sorafenib failure; sorafenib intolerant; Nexavar; Nexavar failure; JX594; oncolytic virus; vaccinia; viral therapy; JX; Biotherapeutics; HEP018; traverse; biologic; Pexa-Vec
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Neoplasms; Vaccinia; Oculocerebral hypopigmentation syndrome type Preus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A (Experimental): Patients on Arm A will receive 1 e9 pfu (plaque forming units) total dose of JX-594 (Vaccinia GM-CSF / TK-deactivated Virus) on each of six (6) treatments over 18 weeks.
  Interventions: Biological: JX-594 recombinant vaccina GM-CSF
- Arm B (Other): Patients on the control arm (Arm B) will have best supportive care over 18 weeks.
  Interventions: Other: Best Supportive Care

INTERVENTIONS:
Biological: JX-594 recombinant vaccina GM-CSF — Patients will be randomised 2:1 to Arm A or Arm B and will receive 6 treatments on days 1, 8, 22, week 6, week 12, and week 18 plus best supportive care as needed.
  Arms: Arm A
Other: Best Supportive Care — Patients will be randomised 2:1 to Arm A or Arm B and will receive best supportive care as needed.
  Arms: Arm B

SUMMARY:
This study is to determine whether JX-594 (Pexa-Vec) plus best supportive care is more effective in improving survival than best supportive care in patients with advanced Hepatocellular Carcinoma (HCC) who have failed sorafenib.

ELIGIBILITY:
KEY Inclusion Criteria:

* Diagnosis of primary HCC by tissue biopsy (histological/cytological diagnosis), or clinical diagnosis
* Previously treated with sorafenib for ≥ 14 days and has discontinued sorafenib treatment at least 14 days prior to randomization due to either intolerance or radiographic progression NOTE: Sorafenib is NOT required to be the most recent treatment received for HCC
* ECOG performance status 0, 1 or 2
* Child-Pugh Class A; or Child-Pugh Class B7 without clinically significant ascites
* Hematocrit ≥30% or Hemoglobin ≥10 g/dL
* Tumor status: Measurable viable tumor in the liver and injectable under imaging-guidance; At least one tumor in the liver that has not received prior local-regional treatment OR that has exhibited >25% growth in viable tumor size since prior local-regional treatment.

KEY Exclusion Criteria:

* Received sorafenib within 14 days prior to randomization
* Received systemic anti-cancer therapy other than sorafenib within 28 days of randomization
* Prior treatment with JX-594
* Platelet count < 50,000 PLT/ mm3
* Total white blood cell count < 2,000 cells/mm3
* Prior or planned organ transplant
* Known significant immunodeficiency due to underlying illness (e.g. HIV/AIDS) and/or medication
* Severe or unstable cardiac disease
* Viable CNS malignancy associated with clinical symptoms
* Pregnant or nursing an infant
* History of inflammatory skin condition (e.g., eczema requiring previous treatment, atopic dermatitis)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2008-12; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Survival | CT scan every six weeks until progression or death, assessed up to 21 months
  Determine overall survival for patients receiving JX-594 plus best supportive care (Arm A) compared with those patients receiving best supportive care (Arm B) in patients with advanced hepatocellular carcinoma (HCC) who have failed sorafenib treatment.

SECONDARY OUTCOMES:
Time to Tumor Progression | CT scan every six weeks until progression or death, assessed up to 21 months
  Determine time-to-tumor-progression (TTP) for Arm A compared with Arm B based on mRECIST for HCC.
Quality of Life | assessed up to 21 months (average)
  Determine the Quality of Life (QoL) of patients treated in Arm A compared with Arm B.
Tumor Response | CT scan every 6 weeks until progression or death, assessed up to 21 months (average)
  Determine tumor response based on mRECIST for HCC of Arm A versus Arm B
Safety profile of JX594 | assessed up to 21 months (average)
  Safety will be assessed by the number of adverse events (AEs) and serious adverse events (SAEs)
Time-to-symptomatic-progression | assessed up to 21 months (average)
  Determine time to progression of Arm A compared to Arm B.

CONTACTS AND LOCATIONS:
Overall Officials: James Burke, MD, Study Director — Jennerex Biotherapeutics
Locations (38):
- United States (11):
  - Moores University of California San Diego Cancer Center, La Jolla, California
  - Chao Family Comprehensive Cancer Center, Orange, California
  - California Pacific Medical Center, San Francisco, California
  - Stanford Hospital and Clinics, Stanford, California
  - University of Chicago Medical Center, Chicago, Illinois
  - Billings Clinic, Billings, Montana
  - Saint Joseph's Hospital, Paterson, New Jersey
  - Montefiore Medical Center, The Bronx, New York
  - Gabrail Cancer Center, Canton, Ohio
  - University Hospitals Case Medical Center, Cleveland, Ohio
  - The Methodist Hospital Department of Surgery, Houston, Texas
- Canada (4):
  - University of Alberta, Edmonton, Alberta
  - University of British Columbia, Vancouver, British Columbia
  - Juravinski Cancer Centre, Hamilton, Ontario
  - Ottawa Hopsital Research Institute, Ottawa, Ontario
- France (6):
  - Hôpitaux Universitaires de Strasbourg - Hôpital Civil, Strasbourg, Alsace
  - Centre Hospitalier Universitaire Hôpital Saint André, Bordeaux, Aquitaine
  - Hôpital de la Croix Rousse, Lyon, Auvergne-Rhône-Alpes
  - CHU d'Estaing, Clermont-Ferrand, Auvergne
  - Hôpital Purpan, Toulouse, Midi-Pyrenees
  - Hôpital Saint Antoine, CPP Ile de France V, Paris, Île-de-France Region
- Germany (4):
  - Klinikum Rechts der Isar der Technischen Universität München, München, Bavaria
  - Medizinische Hochschule Hannover, Hanover, Lower Saxony
  - Johannes Gutenberg-Universität Mainz, Mainz, Rhineland-Palatinate
  - Universitätsklinikum Hamburg-Eppendorf, Hamburg
- Queen Mary Hospital, Hong Kong, Hong Kong
- South Korea (9):
  - Korea University Ansan Hospital, Ansan-si, Gyeonggi-do
  - Kyungpook National University Hospital, Daegu
  - Pusan National University Hospital, Pusan
  - Asan Medical Center, Seoul
  - Korea University Guro Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Seoul National University Hospital, Seoul
  - Severance Hospital,Yonsei University Health System, Seoul
  - Pusan National University Yangsan Hospital, Yangsan
- Taiwan (3):
  - National Cheng-Kung University Hospital, Taipei
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei

REFERENCES:
- [Derived] Moehler M, Heo J, Lee HC, Tak WY, Chao Y, Paik SW, Yim HJ, Byun KS, Baron A, Ungerechts G, Jonker D, Ruo L, Cho M, Kaubisch A, Wege H, Merle P, Ebert O, Habersetzer F, Blanc JF, Rosmorduc O, Lencioni R, Patt R, Leen AM, Foerster F, Homerin M, Stojkowitz N, Lusky M, Limacher JM, Hennequi M, Gaspar N, McFadden B, De Silva N, Shen D, Pelusio A, Kirn DH, Breitbach CJ, Burke JM. Vaccinia-based oncolytic immunotherapy Pexastimogene Devacirepvec in patients with advanced hepatocellular carcinoma after sorafenib failure: a randomized multicenter Phase IIb trial (TRAVERSE). Oncoimmunology. 2019 Jun 3;8(8):1615817. doi: 10.1080/2162402X.2019.1615817. eCollection 2019. PMID 31413923
- See also: Sponsor Website — http://www.jennerex.com